CLINICAL TRIAL: NCT07032805
Title: Telemedicine in Personalized Home Rehabilitation Following Total Knee Arthroplasty (TKA): a Pilot Study
Brief Title: Pilot Study on Personalized Total Knee Arthroplasty (TKA) Rehabilitation Using Telemedicine and Psychoeducation
Acronym: TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Belinda Rizzo (Other)
Collaborators: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Sponsor-Investigator, Laura Belinda Rizzo, Principal Investigator, University of Bari Aldo Moro
Organization: University of Bari Aldo Moro (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prot.2114/CEL
Record Dates: First submitted 2025-05-05; First posted 2025-06-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Arthrosis of the Knee
Keywords: telemedicine; primary osteoarthritis; rehabilitation; posturographic assessment; discontinuation of walking aids; Reduction of pain; physical function; psycho-behavioral assessments; attitude toward technology; use of analgesics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- outpatient rehabilitative treatment plus tele-rehabilitation (Experimental): The study group, after medical, physiotherapeutic, and psychological assessment, will undergo a posturographic exam. They will then receive a treatment focused on strengthening lower limb muscles, improving joint range of motion, enhancing balance, and developing walking ability. This will be delivered in two daily physiotherapy sessions, each lasting 45 minutes, over the 22-25 days of hospitalization. After discharge, they will continue outpatient treatment with two 45-minute sessions per week for three months at a physiotherapy clinic. Additionally, they will receive home supervision from a physiotherapist via telemedicine (video calls using Zoom with encryption), trained on the patient's initial issues identified through posturography and psychological evaluation.
  Interventions: Procedure: personalized outpatient rehabilitation treatment after TKA
- Standard outpatient rehabilitative treatment (Active Comparator): The control group, after medical, physiotherapeutic, and psychological assessments, will undergo a posturographic examination. They will then receive treatment focused on strengthening lower limb muscles, improving joint range of motion, enhancing balance, and gait training. This will be administered in two physiotherapy sessions per day, each lasting 45 minutes, over the 22-25 days of hospitalization. After discharge, they will continue with outpatient physiotherapy consisting of two 45-minute sessions per week for three months at an outpatient physiotherapy clinic.
  Interventions: Procedure: standard outpatient rehabilitation treatment after TKA

INTERVENTIONS:
Procedure: personalized outpatient rehabilitation treatment after TKA — personalized outpatients rehabilitation treatment after TKA, including posturographic assessment, psychomotivational framing, and telemedicine-based rehabilitation interventions
  Arms: outpatient rehabilitative treatment plus tele-rehabilitation
Procedure: standard outpatient rehabilitation treatment after TKA — standard outpatient rehabilitation treatment after TKA
  Arms: Standard outpatient rehabilitative treatment

SUMMARY:
The objective of this clinical trial is to assess the effectiveness of a telemedicine approach in improving treatment adherence and functional outcomes in patients who have recently undergone total knee arthroplasty for primary osteoarthritis. The study focuses on patients aged between 50 and 75 years, with a BMI less than 35, and without known oncological or neurological diseases. Participants will receive personalized rehabilitation treatment, including posturographic assessment, psychomotivational framing, and telemedicine-based rehabilitation interventions. The aim is to provide a framework for adopting more detailed and personalized rehabilitative strategies.

The main research questions are: • Primary: Reduction of pain (VAS), physical function (WOMAC, KOOS). • Secondary: Activities of daily living (Barthel Index, mRS); psycho-behavioral assessments (CEQ, PAM13, CG-PAM, COP-NIV); attitude toward technology (TAM); use of analgesics and walking aids.

Sample size is estimated at 40 patients (20 per group), accounting for a 20% dropout rate, divided into: • Control Group: Standard outpatient rehabilitative treatment with a personalized exercise program. • Study Group: Standard outpatient rehabilitative treatment with a personalized exercise program plus telemonitoring via video calls.

Procedures: • Recruitment and signing of informed consent; • Initial assessment (demographics, baseline tests, and posturography) and initiation of post-acute rehabilitation during hospitalization at T0; • Outpatient rehabilitative interventions with/without tele-rehabilitation support (twice weekly) at discharge, with follow-up assessments at T1 (1.5 months) and T2 (3 months); • Weekly recording of analgesic consumption via a dedicated diary; • Recording the date of discontinuation of walking aids.

DETAILED DESCRIPTION:
To ensure quality and ethical standards in the design and implementation of our randomized clinical trial (RCT), we will apply the Helsinki criteria and the CONSORT checklist. All patients hospitalized for rehabilitation after total knee arthroplasty (TKA) at the San Giovanni di Dio Rehabilitation Center in Adelfia (BA) will be evaluated for eligibility to participate in a clinical study on primary symptomatic osteoarthritis (OA) of the knee between February and May 2025.

Inclusion criteria (in addition to those already mentioned in the brief summary):

Ability to stand on one leg.

Exclusion criteria:

Post-traumatic or inflammatory knee OA. Valgus/varus deformity (hip-knee-ankle angle > or < 10°). The control group and the study group, after medical, physiotherapeutic, and psychological assessment, will undergo a posturographic examination and will then receive a treatment focused on strengthening lower limb muscles, improving joint range of motion, enhancing balance, and gait training. This will be delivered in two physiotherapy sessions per day, each lasting 45 minutes, during the 22-25 days of hospitalization.

Following discharge, participants will receive outpatient treatment consisting of two 45-minute sessions per week for three months at a physiotherapy clinic. The control group will follow this program as usual, while the study group will have the same program reinforced with home supervision via telemedicine. A physiotherapist, trained on the initial posturography findings and psychological assessments, will conduct teleconsultations using Zoom (with end-to-end encryption).

Patient characteristics and outcome measures will be reported in aggregate form, as mean ± standard deviation for continuous variables and absolute frequencies (percentages) for categorical variables. Statistical analysis of outcomes will include testing the significance of differences. The two groups will be compared based on baseline characteristics and changes in outcomes.

The Wilcoxon signed-rank test will be used to evaluate intra-group differences and the effects of the physiotherapy program. The Mann-Whitney U test will be employed to assess differences between groups and evaluate the effect of tele-rehabilitation. The chi-square (χ²) test will be used to verify the homogeneity of categorical variable distributions across the two groups. Statistical significance will be set at p < 0.05. The effect size (ES) for the Mann-Whitney U test will be calculated in the case of between-group comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Recent unilateral total knee arthroplasty;
* Body Mass Index (BMI) < 35;
* Ability to stand on one leg;
* Absence of active known neurological or oncological diseases.

Exclusion Criteria:

* Post-traumatic or inflammatory knee osteoarthritis (OA);
* Valgus/varus deformity (hip-knee-ankle angle > or < 10°).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
VAS (Pain assessment) | At baseline (T0), at 1.5 months (T1), and at 3 months (T2)
  We will use the VAS (Visual Analogue Scale) to quickly and reliably determine the pain perceived by the patient. The VAS (Visual Analogue Scale) consists of a horizontal line 10 centimeters long, with two endpoints representing opposite levels of sensation. Zero is at the extreme left, indicating "No pain," and ten is at the extreme right, representing "The worst pain imaginable." The patient subjectively expresses their perception of pain by indicating a point on the line.
Western Ontario and McMaster Universities Arthritis Index (Physical function) | At baseline (T0), at 1.5 months (T1), and at 3 months (T2)
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a patient-reported outcome questionnaire that assesses symptoms and activity limitations in osteoarthritis or following joint replacement surgery. It evaluates the severity of pain, joint stiffness, and physical function with 24 questions, each using a Likert scale ranging from 0 (no symptoms) to 4 (high intensity or difficulty);
Knee Injury and Osteoarthritis Outcome Score (Knee function) | At baseline (T0), at 1.5 months (T1), and at 3 months (T2)
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-administered questionnaire that assesses symptoms related to the knee joint in osteoarthritis and after total knee replacement surgery. The scale consists of 42 items that evaluate symptoms, pain, daily life functions and activities, sports and recreational activities, and quality of life related to the knee. Responses are on a 5-point Likert scale ranging from 0 (no problems or difficulties) to 4 (severe problems or difficulties).

SECONDARY OUTCOMES:
Barthel Index (Activities of daily living) | At baseline (T0), at 1.5 months (T1), and at 3 months (T2)
  The Barthel Index (BI) for Activities of Daily Living is an ordinal scale that measures a person's ability to perform daily activities through 10 items. Each item is rated by the evaluator based on the individual's capacity to complete the task independently, with assistance, or not at all, with scores as follows:0=unable, 1=needs assistance, 2=independent. The total scores are on a scale from 0 to 100. Interpretation of dependency levels: 0 to 20: Total dependence/21 to 60:Severe dependence/61 to 90:Moderate dependence/91 to 99:Slight dependence.
Modified Rankin Scale (Degree of disability in daily activities) | At baseline (T0), at 1.5 months (T1), and at 3 months (T2)
  The Modified Rankin Scale (mRS) measures the degree of disability, scored from 0 to 6: 0:No symptoms/1:No significant disability despite symptoms/2:Slight disability; unable to perform all previous activities but able to manage own affairs without assistance/3:Moderate disability; requires some help but can walk without assistance/4:Moderately severe disability/5:bedridden, incontinent, and requiring constant care and assistance/6: Dead
Credibility/Expectancy Questionnaire (psychological and behavioral assessment) | At baseline (T0)
  The Credibility/Expectancy Questionnaire(CEQ)measures treatment expectancy and the credibility.It assesses two aspects:cognitive aspects as the reliability of the treatment and emotional aspects, as the belief in improvement related to the treatment.
Patient Activation Measure (Patient activation in managing their illness) | At baseline (T0)
  The Patient Activation Measure (PAM13) evaluates patients' confidence in managing their health condition. It consists of 13 items on a 5point Likert scale:1:Strongly Disagree/2:Disagree/3:Agree/4:Strongly Agree/5:Not Applicable. Scores are converted to a total score ranging from 0 to 100 with four activation levels:1:role is important/2:confidence and knowledge to take action/3:actively taking action/4:maintaining behaviors under stress.
Caregiver/Activation Scale (Caregiver activation) | At baseline (T0)
  The Caregiver/Activation Scale(CG-PAM)is a repeat of the PAM13 and has the same interpretation. It consists of 13 items on a 5point Likert scale:1:Strongly Disagree/2:Disagree/3:Agree/4:Strongly Agree/5:Not Applicable. Scores are converted to a total score ranging from 0 to 100 with four activation levels:1:role is important/2:confidence and knowledge to take action/3:actively taking action/4:maintaining behaviors under stress.
COPing Orientation to Problems Experienced-Italian Version (Assessment of coping styles) | At baseline (T0)
  The COPing Orientation to Problems Experienced-Italian Version(COP-NIV)explores five main independent dimensions. It consists of 60 items assessing how individuals react to stressful events, rated on a 4point scale
Technology Acceptance Model (Technological attitude) | At baseline (T0)
  The Technology Acceptance Model (TAM): consists of 12 items, with six items measuring Perceived Usefulness (PU) and six items measuring Perceived Ease of Use (PEU). PU reflects the degree to which a person believes that using a technology will enhance their job performance, while PEU measures how easy a person believes the technology will be to use. The questions are measured on a Likert-type scale.

OTHER OUTCOMES:
Analgesia | At 1.5 months (T1) and at 3 months (T2)
  Each patient must complete a diary in which they will record their daily consumption of any analgesic medications taken for knee pain throughout the study period, from start to finish. They will report the total consumption weekly and monthly (over 12 weeks / 3 months) and specify the type of medication (paracetamol/NSAIDs/corticosteroids/opioids/muscle relaxants).
Abandonment of mobility aids | At 1.5 months (T1) and at 3 months (T2)
  the complete discontinuation of any prescribed mobility aids will be documented.
Demographic indicators | At baseline (T0)
  age, gender, education level, marital status, employment status, presence of a caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Megna, Professor, Study Director — University Bari "A. Moro"; Teresa Paolucci, Research, Study Director — University of Chieti-Pescara "G. D'Annunzio"; Laura B Rizzo, MD, Principal Investigator — University of Bari "A. Moro"
Locations (1):
- Presidio territoriale di recupero e riabilitazione funzionale "San Giovanni di Dio" Conssi welfare, Adelfia, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT07032805/Prot_SAP_000.pdf